CLINICAL TRIAL: NCT01144793
Title: A Pilot/Observational Study Using a Biomarker Monitoring System to Evaluate Protein Profiles of Neutropenic Fever/Infection in Patients With Acute or Chronic Leukemias Undergoing Chemotherapy or Other Biologic Treatment
Brief Title: Biomarker To Evaluate Protein Profiles of Neutropenic Fever/Infection With Acute or Chronic Leukemias
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Theranos, Inc. (Industry)
Responsible Party: Principal Investigator, Jason Robert Gotlib, Professor of Medicine, Stanford University
Other Study IDs: HEM0008; 98712 (Other: Stanford University Alternate IRB Approval Number); SU-07102008-1246 (Other: Stanford University); 12769 (Other: Stanford IRB)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Leukemia, Lymphocytic; Leukemia, Myeloid
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure, in pilot/observational study, panels of circulating proteins in real time at the onset of neutropenic fever/infection in patients with acute or chronic leukemias undergoing chemotherapy or other biologic treatment. And to generate preliminary trend results in panels of circulating proteins longitudinally during the period of neutropenia and to correlate those values to clinical/laboratory data and patient outcomes.

DETAILED DESCRIPTION:
To identify potential biomarkers for the prediction of NF, we performed serial measurements of nine biomarkers [C-reactive protein (CRP), protein C, interleukin (IL)-6, IL-8, IL-10, IL-1β, tumor necrosis factor-α, monocyte chemotactic protein-1, and intercellular adhesion molecule-1] using a multiplex ELISA array platform every 6-8 hours in patients undergoing myelosuppressive chemotherapy for hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:- Age >= 18

* Pre-admission (ATU, ITA) or inpatient status
* absolute neutrophil count (ANC) <= 1500/mm^3
* Patients with acute myeloid or lymphoid leukemia who:

  * are admitted with newly diagnosed disease and have not yet received induction chemotherapy
  * are admitted with neutropenic fever after receiving post-remission chemotherapy or are admitted for post-remission chemotherapy
* Patients with chronic myeloid leukemia or a chronic lymphoid leukemia/disorder who have received chemotherapy or other disease-specific treatment in the last 30 days where the ANC of <=1500/mm3 is considered by the treating physician to be at least possibly treatment-related
* An intravenous line or catheter (Hickman, port, portacath, or peripherally inserted central venous catheter [PICC] line) must be in place at the time of protocol participation/study start, but will not be inserted solely for the purposes of the study.
* Whenever possible, patients will be consented and blood monitoring will be initiated before the first dose of antibiotic, but if not possible, at no time will standard of care measures will be delayed or interrupted for the purposes of study enrollment.
* Patients must be able to understand the nature of the study and give written informed consent.

There are no exclusion criteria. Anyone who does not meet inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute or Chronic Leukemias
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robert Gotlib, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan SM, Chadwick J, Young DL, Holmes E, Gotlib J. Intensive serial biomarker profiling for the prediction of neutropenic Fever in patients with hematologic malignancies undergoing chemotherapy: a pilot study. Hematol Rep. 2014 Jun 23;6(2):5466. doi: 10.4081/hr.2014.5466. eCollection 2014 Apr 22. PMID 25013718